CLINICAL TRIAL: NCT06968013
Title: Investigating on the Efficacy of Well-Being Therapy (WBT) for Chronic Insomnia (CI) With Depressive Symptoms
Brief Title: Effect of WBT for CI With Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBT-CI-D-2025
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Chronic Insomnia; Depression Disorders
Keywords: Chronic Insomnia; Depression Disorders; Well-Being Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WBT-CI (Experimental)
  Interventions: Behavioral: Well-Being Therapy
- SHE-CI (Active Comparator)
  Interventions: Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Behavioral: Well-Being Therapy — Participants will undergo Well-Being Therapy (WBT) sessions once daily for 50 minutes over a period of six weeks. The core elements of WBT include prompting participants to identify instances of well-being, contextualize these experiences using a structured diary, and recognize as well as restructure thoughts, beliefs, and behaviors that prematurely disrupt well-being. Additionally, the specific components of the six dimensions of the Psychological Well-Being (PWB) scale-autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance-are systematically integrated into different therapy sessions
  Arms: WBT-CI
Behavioral: Sleep Hygiene Education — Participants will receive Sleep Hygiene Education (SHE) alone for 6 weeks. SHE involves education on maintaining consistent sleep schedules, creating a sleep-conducive environment, reducing stimulant use (e.g., caffeine, alcohol), and promoting healthy daily routines to improve sleep quality.
  Arms: SHE-CI

SUMMARY:
This randomized controlled trial aims to explore the therapeutic effects of Well-Being Therapy (WBT) on patients with Chronic Insomnia accompanied by depressive symptoms.

DETAILED DESCRIPTION:
According to DSM-IV criteria, approximately 6%-10% of the adult population in industrialized countries suffer from chronic insomnia (CI), characterized by difficulties in initiating or maintaining sleep accompanied by daytime symptoms persisting for at least four weeks. Chronic insomnia often leads to various psychiatric symptoms, with depressive symptoms being among the most common. For patients with CI and comorbid depressive symptoms, the most common treatment involves the use of antidepressant medications. However, while depressive symptoms may improve, insomnia symptoms often persist.

Among non-pharmacological interventions aimed at promoting psychological well-being, Well-Being Therapy (WBT) stands out as a brief and innovative psychotherapeutic approach. WBT is a structured, manualized, short-term therapy that incorporates self-monitoring of well-being episodes through the use of a diary, cognitive restructuring of interfering thoughts and behaviors, and homework assignments.

Previous research has demonstrated the effectiveness of WBT in alleviating stress in populations experiencing 'allostatic load.' This study seeks to evaluate the therapeutic effects of six WBT sessions on individuals with CI and comorbid depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Insomnia Disorder according to DSM-5 criteria, with a duration of at least 3 months.
2. Pittsburgh Sleep Quality Index (PSQI) total score > 5.
3. Age 8 years or older.
4. Educational level of at least junior high school.
5. Voluntarily agree to participate and provide written informed consent.
6. Presence of depressive symptoms, defined as Hamilton Depression Scale (HAMD) score ≥ 16.

Exclusion Criteria:

1. Presence of severe physical illnesses or major psychiatric disorders, or at risk of suicide.
2. Diagnosed or suspected of having sleep breathing disorders, restless legs syndrome, circadian rhythm sleep disorders, or engaged in shift work.
3. Pregnant or breastfeeding women.
4. Currently undergoing any psychological therapy.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) Score at 6 Weeks | Baseline and Week 6
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire designed to evaluate sleep quality over a one-month period. It consists of 19 items grouped into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each component is scored on a scale of 0 to 3, and the total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.

SECONDARY OUTCOMES:
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) Scores at 3, 6, and 12 Months | Baseline, 3 months, 6 months, and 12 months
  As mentioned in the previous text.
Change from Baseline in Hamilton Depression Scale-17 (HAMD-17) Scores | Baseline, Week 6, 3 months, 6 months, and 12 months
  The Hamilton Depression Scale-17 (HAMD-17) is a clinician-administered tool designed to assess the severity of depressive symptoms over the past week. It consists of 17 items that evaluate various aspects of depression, such as mood, guilt, insomnia, anxiety, and physical symptoms. Each item is scored on a scale, and the total score reflects the severity of depression.
  The scoring criteria are as follows:
  0-7: Normal (not depressed) 8-13: Mild depression 14-18: Moderate depression 19-22: Severe depression 23 or above: Very severe depression.
Change from Baseline in Beck Depression Inventory-II (BDI-II) Scores | Baseline, Week 6, 3 months, 6 months, and 12 months
  The Beck Depression Inventory-II (BDI-II) is a self-report questionnaire designed to assess the severity of depressive symptoms. It consists of 21 items, each scored on a scale from 0 to 3, with a total score ranging from 0 to 63. The scoring interpretation is as follows:
  0-13: Minimal depression 14-19: Mild depression 20-28: Moderate depression 29-63: Severe depression
Change from Baseline in Beck Anxiety Inventory (BAI) Scores | Baseline, Week 6, 3 months, 6 months, and 12 months
  The scale contains 21 items and uses a 4-point scale method, with a total score of 15-25 as mild anxiety, 26-35 as moderate anxiety, and 36 or more as severe anxiety
Change from Baseline in Patient Health Questionnaire-4 (PHQ-4) Scores | Baseline, Week 6, 3 months, 6 months, and 12 months
  The Patient Health Questionnaire-4 (PHQ-4) is a brief screening tool designed to assess symptoms of anxiety and depression. It consists of four items, with two questions focusing on anxiety and two on depression. Each item is scored from 0 to 3, resulting in a total score ranging from 0 to 12. The scoring interpretation is as follows:
  0-2: None (minimal distress) 3-5: Mild distress 6-8: Moderate distress 9-12: Severe distress
Change from Baseline in 36-Item Short Form Health Survey (SF-36) Scores | Baseline, Week 6, 3 months, 6 months, and 12 months
  The 36-Item Short Form Health Survey (SF-36) is a widely used questionnaire designed to measure health-related quality of life. It evaluates eight domains: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each domain is scored on a scale from 0 to 100, with higher scores indicating better health status.
Change from Snaith-Hamilton Pleasure Scale (SHAPS) Scores | Baseline, Week 6, 3 months, 6 months, and 12 months
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a self-report questionnaire designed to measure anhedonia, which is the reduced ability to experience pleasure. It consists of 14 items assessing various aspects of enjoyment in daily life, such as hobbies, social interactions, and sensory experiences. Each item is scored on a scale, and the total score ranges from 0 to 14, with higher scores indicating greater levels of anhedonia.
Change from Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) Scores | Baseline, Week 6, 3 months, 6 months, and 12 months
  The Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) is a self-report questionnaire designed to assess maladaptive beliefs and attitudes related to sleep. It consists of items scored on a scale, typically using a visual analogue format or numerical ratings. The total score is calculated by averaging responses across all items, with higher scores indicating more dysfunctional beliefs about sleep.
Change from Insomnia Severity Index (ISI) Scores | Baseline, Week 6, 3 months, 6 months, and 12 months
  The scale is divided into 7 sections with a total score of 0-28, with higher scores indicating more severe insomnia. The degree of insomnia is classified according to the scores: 0-7 indicates no insomnia, 8-14 is mild insomnia, 15-21 is moderate insomnia, and 22-28 is severe insomnia.
Change in Self-rated Sleep Severity (0-10 Numeric Rating Scale) | Baseline, Week 6, 3 months, 6 months, and 12 months
  The Self-rated Sleep Severity (0-10 Numeric Rating Scale) is a simple tool used to assess an individual's perception of their sleep quality or severity of sleep-related issues. Respondents rate their sleep on a scale from 0 to 10, where 0 represents no sleep problems and 10 indicates the most severe sleep difficulties.
Frequency and Severity of Adverse Events | Throughout study duration up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu X, Song P, Yin L, Wang K, Zhu B, Huang X, Niu Y, Leng H, Xue Q, Peng M, Min B, Shangguan F, Zhang P, Zhao W, Wang H, Lv J, Yang M, Wang P, Li D, Gao X, Feng K, Yun K, Cosci F, Wang H. The Role of Online Well-Being Therapy in Overcoming Allostatic Overload in Medical Workers: A Pilot Randomized Controlled Study. Psychother Psychosom. 2024;93(5):316-327. doi: 10.1159/000540924. Epub 2024 Sep 23. PMID 39312891